CLINICAL TRIAL: NCT02526875
Title: A Multicenter, Prospective, Randomized, Open-label, Phase 4 Trial Designed to Evaluate the Efficacy of a Telmisartan/S-Amlodipine(Telminuvo®Tab. 40/2.5mg) on 24-hour BP Control in Hypertensive Patients Inadequately Controlled
Brief Title: Efficacy of a Telmisartan/S-Amlodipine on 24-hour BP Control in Hypertensive Patients Inadequately Controlled
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 330HT14009
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: hypertension, Telmisartan/S-Amlodipine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- night (Experimental): Telminuvo®Tab. 40/2.5mg ,Once daily, from 6 pm to 10 pm, Per oral for 8weeks after 2~4weeks run-in period with Telmitrend®Tab. 40mg
  Interventions: Drug: Telminuvo®Tab. 40/2.5mg
- morning (Active Comparator): Telminuvo®Tab. 40/2.5mg ,Once daily, from 6 am to 10 am, Per oral for 8weeks after 2~4weeks run-in period with Telmitrend®Tab. 40mg
  Interventions: Drug: Telminuvo®Tab. 40/2.5mg

INTERVENTIONS:
Drug: Telminuvo®Tab. 40/2.5mg — per oral for 8weeks after 2~4weeks run-in period with Telmitrend®Tab. 40mg
  Other Names: Telmisartan/S-Amlodipine 40/2.5mg

SUMMARY:
To Evaluate the Efficacy of the Timing of the Administration of a Telmisartan/S-Amlodipine (Telminuvo®Tab. 40/2.5mg) on 24-hour BP Control in Hypertensive Patients Inadequately Controlled by Telmisartan Monotherapy

DETAILED DESCRIPTION:
A Multicenter, Prospective, Randomized, Open-label, Phase 4 Trial Designed to Evaluate the Efficacy of the Timing of the Administration of a Telmisartan/S-Amlodipine(Telminuvo®Tab. 40/2.5mg) on 24-hour BP Control in Hypertensive Patients Inadequately Controlled by Telmisartan Monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. More than 20 years in hypertension patient
2. Hypertension is satisfied with the Clinic blood pressure that was measured at the time of screening

   * Treatment-Naive: Clinic Mean sitting diastolic blood pressure ≥ 100mmHg.
   * Treatment-Experienced: Clinic Mean sitting diastolic blood pressure ≥ 90mmHg.
3. Hypertension is satisfied with the Clinic blood pressure that was measured at the time of randomization

   * Clinic Mean sitting diastolic blood pressure ≥ 90mmHg
4. Patient who decided to participate and signed on an informed consent form willingly

Exclusion Criteria:

1. Clinic Mean sitting systolic blood pressure ≥ 180mmHg or Clinic Mean sitting diastolic blood pressure ≥ 115mmHg at the time of Screening and Randomization
2. As night workers who sleep during the day and whose working hours including 00:00 to 04:00
3. Secondary Hypertension
4. Severe heart disease(Heart failure; New York Heart Association(NYHA) class 3, 4) and recent unstable angina or myocardial infarction or valvular heart disease or arrhythmia requiring treatment within the past 3 months
5. Severe cerebrovascular disorders such as cerebral infarction, cerebral hemorrhage within 6 months
6. type 1 diabetes mellitus or Uncontrolled type 2 diabetes mellitus(HbA1c > 8.0%)
7. Severe or malignant retinopathy
8. Abnormal laboratory test results

   * Aspartate aminotransferase/Alanine aminotransferase > Upper normal limit X 2
   * Serum creatinine > Upper normal limit X 2
9. Acute of chronic inflammatory status requiring treatment
10. Need for other antihypertensive drugs during the trial
11. Need for prohibited medication specified in the protocol
12. A history of angioedema with ACE inhibitors or angiotensin-Ⅱ receptor blockers
13. Severe hypersensitivity to amlodipine or telmisartan
14. History of drug or alcohol abuse within 6 months
15. Surgical or medical conditions

    * History of major gastrointestinal surgery
    * History of active inflammatory bowel syndrome within 12 months
    * Abnormal pancreatic functions
    * Gastrointestinal/rectal bleeding
    * Urinary tract obstruction
16. Administration of other Investigational Product within 30 days
17. Pregnant, breast-feeding and childbearing age who don't use adequate contraception
18. History of malignant tumor within 5 years (including leukemia and lymphoma)
19. Another clinical condition in investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the 24hr mean blood pressure by ambulatory blood pressure monitoring(ABPM) at week 8. | Baseline and week 8
  Change from baseline in the 24hr mean blood pressure by ambulatory blood pressure monitoring(ABPM) at week 8.

SECONDARY OUTCOMES:
Change from baseline in the 24hr mean daytime, nighttime, morning blood pressure by ABPM at week 8 | Baseline and week 8
  * Daytime: 06:00~21:59
  * Nighttime: 22:00~05:59
  * Morning: 06:00~11:59
Change from baseline in the clinic mean blood pressure at week 8. | Baseline and week 8
24hr ABPM and Clinic BP control at week 8. | Baseline and week 8
  <24hr ABPM>
  * 24hr mean BP: 24hr mean Systolic blood pressure(SBP)<130mmHg and 24hr mean Diastolic blood pressure(DBP)<80mmHg
  * Daytime BP: Daytime mean SBP<135mmHg and Daytime mean DBP<85mmHg
  * Night time BP: Night time mean SBP<120mmHg and Night time mean DBP<70mmHg
  <Clinic BP>
  : Mean sitting systolic blood pressure<140mmHg and Mean sitting diastolic blood pressure<90mmHg
Morning BP Surge | Baseline and week 8
  The morning BP surge was calculated as the morning BP minus the lowest BP. Morning BP was defined as the average BP during the first 2 h after waking. The lowest BP was defined as the average of three BP readings focused on the lowest night-time reading (that is, the lowest reading plus the readings immediately before and after)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Gu Shin, Principal Investigator — Yeungnam University Hospital
Locations (10):
- South Korea (10):
  - Korean University Guro Hospital, Seoul, Guro-gu
  - Myongji Hospital, Goyang, Gyeonggi-di
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Bundang Jesaeng Hospital, Seongnam-si, Gyeonggi-do
  - Daegu Catholic University Medical Center, Dae-gu, Gyeongsangbuk-do
  - Keimyung University Dongsan Medical Center, Daegu, Gyeongsangbuk-do
  - Yeungnam University Medical Center, Daegu, Gyeongsangbuk-do
  - Cheju Halla General Hospital, Jeju City, Jeju Special Self-Governing
  - Dong-A University Hospital, Busan, Seo-gu
  - Pusan National University Hospital, Busan, Seo-gu

IPD SHARING:
Plan to Share IPD: No